CLINICAL TRIAL: NCT06432062
Title: Investigation the Effect of Rectus Abdominis and Erector Spinae Muscle Fatigue on the Viscoelastic Properties of Thoracolumbal Fascia
Status: Completed | Type: Observational
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Hatice Karabulut, Principal Investigator, Istanbul Saglik Bilimleri University
Other Study IDs: 2022-13596
Record Dates: First submitted 2024-05-08; First posted 2024-05-29 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Muscle Weakness
Keywords: rectus abdominis; erector spinae; thoracolumbar fascia
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The rectus abdominis, which enables the trunk to flex with its activation, and the erector spinae muscles, which provide trunk extension with its activation, are among the structures located in the core region and involved in the stabilization of the spine. While the muscles in the core area actively provide the stabilization of the medulla spinalis, this stabilization is also supported by passive subsystems. Passive subsystem fascia etc. creates structures. Thoracolumbar fascia is one of the important fascias due to its connections with the muscles in the core area. Fatigue etc. of the structures in the core area. As a result of physiological processes, their functionality may decrease, which may affect the stabilization of the core area. Fatigue occurs as a result of lactic acid accumulation in the structures in the body and this process is called the recovery period. The types of exercises performed also affect the recovery period. For this reason, different exercise types such as dynamic and static can be used when creating exercise programs. Due to the functions of the rectus abdominis and erector spinae muscles and thoracolumbar fascia in the body, their effects on the spine and their connections with each other; It is aimed to examine the effect of muscle fatigue in these muscles on the viscoelastic properties of the thoracolumbar fascia and their recovery rates.

ELIGIBILITY:
Inclusion Criteria:

* Being a healthy individual between the ages of 18-35
* Not having any chronic disease
* Body mass index (BMI) is 24.9 kg/m2 or lower
* Volunteering to participate in the study

Exclusion Criteria:

* Having a chronic illness (Diabetes, blood pressure, etc.)
* Having a diagnosed spine problem
* Being diagnosed with scoliosis
* Pilates, yoga, etc. in the last 6 months. to have done sports
* Beighton score of 4 or above
* Being diagnosed with cardiopulmonary system disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will be conducted with healthy male individuals between the ages of 18-35. Individuals without any orthopedic, neurological or chronic disease will be included in the study.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Thoracolumbal Fascia Viscoelastic Properties | 2 weeks
  Viscoelastic properties of the thoracolumbal fascia (TFL) was performed with the MyotonPRO™ (Myoton AS, Estonia) device. Before and after imeddiately after application of the fatigue protocol. The measurement point determined for TFL of individuals rest were marked with a medical marker pen. During the measurement, the probe of the device was adjusted to pulse once into the skin with a force of 0.4 N and for 15 ms. During the test, the tip of the MyotonPro™ device was placed perpendicular to the marked area and gently pressed against the skin at a depth of 3 mm until the green light came on.

SECONDARY OUTCOMES:
Fatigue Assessment with Borg Scale | 2 weeks
  Fatigue assessment will be made using the Modified Borg Scale. The Modified Borg Scale is a subjective evaluation method that evaluates fatigue and shortness of breath during activity or at rest between 0 and 10. 0 points "not at all" means the lowest, and 10 points "very severe" means the highest fatigue and shortness of breath.
Investigations of Recovery Times | 2 weeks
  Moxy®, (Moxy®, Fortiori Design LLC, Minnesota, USA) Monitor will be used to detect the change in intramuscular oxygen saturation of the muscles and the time it takes to return to resting levels during and after fatigue protocols. The most swollen areas of the rectus abdominis and erector spinae muscles will be marked with a cosmetic pen and the device will be placed.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Health Science University, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No